CLINICAL TRIAL: NCT00001512
Title: Active Specific Immunotherapy for Follicular Lymphomas With Tumor-Derived Immunoglobulin Idiotype Antigen Vaccines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 960133; 96-C-0133; NCT00878488 (obsolete NCT alias)
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-03-05

CONDITIONS: B Cell Lymphoma; Follicular Lymphoma; Lymphoma
Keywords: ProMace Chemotherapy; Indolent Lymphoma; Anti-Idiotype Antibody; GM-CSF; B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Follicular; Lymphoma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

INTERVENTIONS:
Drug: Id-KLH Vaccine
Drug: GM-CSF

SUMMARY:
The idiotype of the immunoglobulin on a given B cell malignancy (Id) can serve as a clonal marker, and a previous pilot study in lymphoma patients has demonstrated that autologous Id protein can be formulated into an immunogenic, tumor specific antigen by conjugation to a carrier protein (KLH) and administration with an emulsion-based adjuvant. The goals of vaccine development in the current study are to develop vaccines: 1) with improved potency and 2) which are more effective at inducing cell-mediated immune responses. The selection of GM-CSF as the immunological "adjuvant" is a direct extension of our laboratory studies in small animal models demonstrating that GM-CSF can enhance the potency of the prototype Id-KLH vaccine by augmenting almost exclusively the cellular arm of the immune response.

The objectives of this study are: 1) to evaluate cellular and humoral immune responses against the unique idiotype of the patient's lymphoma and 2) to evaluate the ability of the Id vaccine to clear the bone marrow of malignant cells detectable by pathologic examination or molecular examination (polymerase chain reaction amplification of the rearranged bcl-2 oncogene).

The goal of this study is to treat previously untreated patients with follicular lymphomas to complete remission or minimal residual disease with ProMACE chemotherapy. Three to six months after completion of chemotherapy, in an effort to reduce the relapse rate (by eradicating microscopic disease resistant to chemotherapy), patients will receive an autologous Id vaccine administered in combination with GM-CSF. Id-KLH (0.5 mg) is administered subcutaneously. GM-CSF is administered subcutaneously locally with the vaccine on the day of vaccination and for the three consecutive days following vaccination as close to the initial vaccination site as possible at one of two doses (patients are randomized to either a high or low dose, 500 or 100 micrograms/m2).

We plan to accrue 42 patients. Twenty-nine patients have been enrolled. Sixteen patients have entered and/or completed the vaccination phase. Patients have demonstrated significant lymphoproliferative responses specific for autologous idiotype of a magnitude which is significantly greater than previously observed.

DETAILED DESCRIPTION:
The idiotype of the immunoglobulin on a given B cell malignancy (Id) can serve as a clonal marker, and a previous pilot study in lymphoma patients has demonstrated that autologous Id protein can be formulated into an immunogenic, tumor specific antigen by conjugation to a carrier protein (KLH) and administration with an emulsion-based adjuvant. The goals of vaccine development in the current study are to develop vaccines: 1) with improved potency and 2) which are more effective at inducing cell-mediated immune responses. The selection of GM-CSF as the immunological "adjuvant" is a direct extension of our laboratory studies in small animal models demonstrating that GM-CSF can enhance the potency of the prototype Id-KLH vaccine by augmenting almost exclusively the cellular arm of the immune response.

The objectives of this study are: 1) to evaluate cellular and humoral immune responses against the unique idiotype of the patient's lymphoma and 2) to evaluate the ability of the Id vaccine to clear the bone marrow of malignant cells detectable by pathologic examination or molecular examination (polymerase chain reaction amplification of the rearranged bcl-2 oncogene).

The goal of this study is to treat previously untreated patients with follicular lymphomas to complete remission or minimal residual disease with ProMACE chemotherapy. Three to six months after completion of chemotherapy, in an effort to reduce the relapse rate (by eradicating microscopic disease resistant to chemotherapy), patients will receive an autologous Id vaccine administered in combination with GM-CSF. Id-KLH (0.5 mg) is administered subcutaneously. GM-CSF is administered subcutaneously locally with the vaccine on the day of vaccination and for the three consecutive days following vaccination as close to the initial vaccination site as possible at one of two doses.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must meet all of the following eligibility criteria.

Tissue diagnosis of: follicular small cleaved cell, or follicular mixed lymphoma with surface IgM, IgG or IgA phenotype with a monoclonal heavy and light chain. Pathology slides must be submitted to the NIH Pathology Department for review.

Stage III or IV lymphoma.

Only previously untreated patients are eligible.

Previous treatment with radiation alone (less than TBI) is permissible.

A single peripheral lymph node of at least 2 cm size accessible for biopsy/harvest.

Karnofsky status greater than or equal to 70 percent.

Life expectancy of greater than 1 year.

Serum creatinine less than or equal to 1.5 mg per dl unless felt to be secondary to lymphoma.

Bilirubin less than or equal to 1.5 mg/dl unless felt to be secondary to lymphoma or Gilbert's disease. SGOT/SGPT less than or equal to 3.5 times upper limit of normal.

Ability to give informed consent. Ability to return to clinic for adequate follow-up for the period that the protocol requires.

EXCLUSION CRITERIA:

Prior total body irradiation.

Presence of antibodies to HIV, hepatitis B surface antigen or other active infectious process.

Pregnancy or lactation. Fertile men and women must plan to use effective contraception. A beta-HCG level will be obtained in women of child-bearing potential.

Patients with previous or concomitant malignancy, regardless of site, except curatively treated squamous or basal cell carcinoma of the skin, or effectively treated carcinoma in situ of the cervix.

Patients unwilling to give informed consent.

Failure to meet any of the inclusion criteria.

Any medical or psychiatric condition that in the opinion of the protocol chairman would compromise the patient's ability to tolerate this treatment will be excluded from this protocol.

Patient with CNS lymphoma (current or previously treated) will not be eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 1996-09-09; Primary Completion 2010-03-05 (Actual); Study Completion 2010-03-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Stevenson GT, Stevenson FK. Antibody to a molecularly-defined antigen confined to a tumour cell surface. Nature. 1975 Apr 24;254(5502):714-6. doi: 10.1038/254714a0. No abstract available. PMID 47617
- [Background] Miller RA, Maloney DG, Warnke R, Levy R. Treatment of B-cell lymphoma with monoclonal anti-idiotype antibody. N Engl J Med. 1982 Mar 4;306(9):517-22. doi: 10.1056/NEJM198203043060906. No abstract available. PMID 6173751
- [Background] Daley MJ, Gebel HM, Lynch RG. Idiotype-specific transplantation resistance to MOPC-315: abrogation by post-immunization thymectomy. J Immunol. 1978 May;120(5):1620-4. PMID 77876